CLINICAL TRIAL: NCT06043635
Title: Predictors of Inhaled Nitric Oxide (iNO) Responsiveness in Neonates With Persistent Pulmonary Hypertension of the Newborn (PPHN)/Hypoxic Respiratory Failure (HRF)
Brief Title: Predictors of Inhaled Nitric Oxide Responsiveness in Patients With PPHN
Acronym: PINOR
Status: Withdrawn | Type: Observational
Why Stopped: No patients were enrolled
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Bernadette Chen, Principal Investigator, Nationwide Children's Hospital
Other Study IDs: IRB18-00711
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: PPHN; Hypoxic Respiratory Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, tracheal aspirate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify biochemical, clinical, or genetic biomarkers that may predict responsiveness to iNO in neonates with PPHN/HRF. The primary outcome will be identification of any biomarker(s) associated with response to iNO therapy. We will evaluate related biomarkers at various time-points during disease progression and in response to therapy, including single nucleotide polymorphisms in the cyclic adenosine monophosphate/cyclic guanosine monophosphate-Phosphodiesterase (PDE) pathway, indicators of metabolic dysregulation and inflammation, as well as biochemical markers of heart strain. We will perform targeted neonatal echocardiograms to evaluate severity of PPHN and heart function both as an added clinical biomarker and to follow disease progression.

DETAILED DESCRIPTION:
A single-center, prospective observational cohort study evaluating potential biochemical, clinical, and/or genetic biomarkers in neonates admitted with a diagnosis of PPHN that may predict iNO response. Thus, it is important to collect data prior to the initiation of iNO to be able to identify biomarkers that can predict response. For patients who meet the screening criteria and when consent is not attainable prior to initiation of the potential life-saving iNO therapy, then samples will be obtained with deferred written informed parental consent obtained within the first 4 hours after enrollment. These patients will have one sample of blood, urine, and tracheal aspirate (if available) collected. If the patient meets the inclusion and exclusion criteria, the patient will be recruited for study participation. To ensure no delay in care or in the initiation of the only FDA-approved vasodilator for this population, iNO, a deferred written informed parental consent is requested to allow for the collection of blood, urine, tracheal aspirate specimens (if available) prior to the initiation of iNO. Only one sample of blood and tracheal aspirate specimens will be collected prior to the deferred consent. Samples are often collected during the routine collections that are obtain from patients who are critically ill such as in our study participants, therefore, no additional discomfort will be expected from this study. Urine collection will be from cotton ball collection that would normally be discarded and is noninvasive. All data and biospecimens obtained from eligible infants whose parent(s) decline consent or do not qualify for the study will be discarded.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 34 weeks gestational age.
2. Less than or equal to 10 postnatal days of age.
3. Echocardiographic evidence of PPHN (right-to-left or bidirectional shunt at the foramen ovale or the ductus arteriosus and/or severe tricuspid regurgitation)

Exclusion Criteria:

1. Lethal congenital anomalies, obvious syndromic or chromosomal disorders.
2. Congenital diaphragmatic hernia.
3. Congenital heart defect (except a small atrial septal defect, ventricular septal defect, and/or PDA).

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Late pre-term and term neonates admitted to NCH NICU with a diagnosis of PPHN/HRF.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Biomarker Identification | 24 hours after enrollment
  Identification of a biomarker that is associated with response to iNO therapy

SECONDARY OUTCOMES:
Biomarker Predication | 24 hours after enrollment
  Identification of a biomarker that may be predictive of the need for iNO therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Chen, MD, Principal Investigator — Nationwide Children's Hospital

IPD SHARING:
Plan to Share IPD: No